CLINICAL TRIAL: NCT04350008
Title: BIO|CONCEPT.Renamic Neo
Brief Title: BIO|CONCEPT.Renamic Neo Study
Status: Completed | Type: Observational
Sponsor: Biotronik Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biotronik SE & Co. KG (Industry)
Other Study IDs: BA112
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2020-05

CONDITIONS: Medical Devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Renamic Neo programmer device, including software; PK-222-L ECG cable — Patients were enrolled either for implantation including subsequent pre-hospital discharge or for a follow-up visit only. ICM patients were included for follow-ups only. Implants were programmed and interrogated by using the investigational devices.

SUMMARY:
The BIO|CONCEPT.Renamic.Neo study is designed as a pre-market study to provide clinical data and supporting evidence of the safety, performance and usability of the Renamic Neo programmer system.

ELIGIBILITY:
Inclusion Criteria:

* Patient is planned for de novo implantation or already has a BIOTRONIK active, implantable device.
* Patient is able to understand the nature of the study and provides written informed consent.

Exclusion Criteria:

* Patient is implanted with a Stratos pacemaker.
* Patient is planned for implant exchange or upgrade.
* Patient is pregnant or breast feeding.
* Patient is less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are planned to receive or are already implanted with a programmable BIOTRONIK cardiac rhythm management (CRM) device.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - GenesisCare Wesley, Auchenflower
  - GenesisCare Bundaberg, Bundaberg
  - The Canberra Hospital, Canberra
  - Lyell McEwin Hospital (LMH), Elizabeth Vale
  - Monash Medical Centre, Melbourne
  - Mulgrave Private Hospital, Mulgrave
  - John Hunter Hospital, New Lambton Heights

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Implantation and Follow-up Use Cases: Implantation use cases including PSA measurements. Pre-hospital discharges of these patients account for follow-up use cases
Period: Overall Study
Arm/Group | Implantation and Follow-up Use Cases
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Implantation and Follow-up Use Cases
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 110
Height [cm] [Mean (Standard Deviation); unit: cm] | 171.4 (10.3)
Weight [kg] [Mean (Standard Deviation); unit: kg] | 84.5 (19.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Device Effects (ADE) and Device Deficiencies (DD) Per Number of Implantations and Per Number of PHD/Follow-up Cases
Description: The number of Adverse Device Effects (ADE) and Device Deficiencies (DD) that occured in patients, users or other persons during the use of the Renamic Neo programmer at implantation, pre-hospital discharge and during the on-site follow-up was evaluated. The investigator was asked to report any ADEs or DD that occurred during implantations and follow-ups. All Adverse Device Effects (ADE) related to the investigational device and only Device Deficiencies (DD) that were determined to bear the potential for a medical occurrence were prespecified to be collected.
Time Frame: Patients participated from (I) implantation until the pre-hospital discharge (usually 1-2 days) or (II) only for the in-office follow-up (usually 1 day).
Population: Analysed were 49 implantation use cases and 102 follow-up use cases which include interrogations at pre-hospital discharge. Analysed were all implantation, pre-hospital discharge and follow-up cases for which the Renamic Neo programmer was used.
Measure: Count of Units; unit: use cases for Renamic Neo
Units Other Than Participants: use cases for Renamic Neo
Groups:
- Implantation and Follow-up Use Cases: Implantation use cases include PSA measurements. Pre-hospital discharges of these patients account for follow-up use cases
Arm/Group | Implantation and Follow-up Use Cases
Number analyzed (Participants) | 110
Number analyzed (use cases for Renamic Neo) | 151
use cases for Renamic Neo | 0

ADVERSE EVENTS:
Time Frame: Implantations (Days): Mean: 1.0; SD: SD:1.6 Follow-up (Days) : Mean:1.1 SD: 6.0
Arm/Group | Implantation and Follow-up Use Cases
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 1/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation and Follow-up Use Cases (N=110)
Complete heart block (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04350008/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04350008/SAP_001.pdf